CLINICAL TRIAL: NCT02844907
Title: Regulation of Insulin Secretion by the GLP-1 Receptor
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding expired
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Durham VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ENDA-006-15S; Pro00070325 (Other: Duke University); 01992 (Other: Durham VA Medical Center)
Record Dates: First submitted 2016-07-22; First posted 2016-07-26 (Estimated); Results first posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-11

CONDITIONS: Insulin Secretion
Keywords: Incretins; GLP-1; Exendin-9; Insulin Resistance; Diabetes; Pre-diabetes
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus; Glucose Intolerance | interventions — exendin (9-39); Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyperglycemic clamp + Exendin (9-39) (Experimental): During the 2-hour procedure, a variable infusion of 20% dextrose and blood glucose will be clamped at basal + 3mM. Participants will receive an infusion of the GLP-1 receptor antagonist Exendin (9-39) between the 60-120 minute time-points of the clamp. The amount of Ex-9 infused will be 750 pmol/kg/min for 60 minutes.
  Interventions: Drug: Exendin (9-39); Other: Hyperglycemic Clamp
- Dexamethasone (Experimental): Subjects will be asked to take 4 mg once daily between Visit-2 and Visit-3.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Exendin (9-39) — Upon establishing a hyperglycemic clamp (target blood glucose at basal +3 mM) Exendin (9-39) will be infused.
  Other Names: GLP-1 receptor antagonist
  Arms: Hyperglycemic clamp + Exendin (9-39)
Drug: Dexamethasone — Between Visit-2 and Visit-3, Dexamethasone (4 mg tablet) once daily for 5-7 days.
  Arms: Dexamethasone
Other: Hyperglycemic Clamp — A variable infusion of 20% dextrose will begin to clamp the blood glucose at basal +3 mM.
  Arms: Hyperglycemic clamp + Exendin (9-39)

SUMMARY:
AIM2: The purpose of Aim-2 of this study is to determine the role of basal GLP-1 action on the beta-cell response to insulin resistance. Healthy subjects will have fasting GLP-1 action determined with GLP-1r blockade before and after induction of experimental insulin resistance. The investigators hypothesize that fasting GLP-1 action will increase to compensate for experimental insulin resistance.

AIM3: The purpose of Aim-3 of this study is to determine the role of basal GLP-1 action on fasting glucose regulation in lean, obese, pre-diabetic and type 2 diabetic (T2DM) subjects. A cross sectional study of age-matched subjects across the spectrum of glucose tolerance will be used to test the hypothesis that fasting GLP-1 action increases as beta-cell function declines.

DETAILED DESCRIPTION:
AIM2: The purpose of this study is to determine the role of basal GLP-1 action on the beta-cell response to insulin resistance. Healthy subjects will have fasting GLP-1 action determined with GLP-1r blockade before and after induction of experimental insulin resistance. The investigators hypothesize that fasting GLP-1 action will increase to compensate for experimental insulin resistance.

The study will enroll up to 20-25 healthy participants and while it is anticipated that the screening blood draw will yield a number of screen failures, it is estimated that 10-15 subjects will complete the entire study protocol. Enrolled participants will be asked to complete three study visits including the consent visit and two infusion study visits that will include hyperglycemic clamp procedures with the addition of the GLP-1 receptor antagonist Exendin (9-39) to determine the fasting GLP-1 effect. Each infusion procedure will last 2 hours. Subjects will be asked to take dexamethasone daily for approximately one week between Visit-2 and Visit-3 to induce insulin resistance.

The investigators will enroll 6-10 additional subjects as controls for effects of time and repeat testing. These individuals will have identical clamps with no dexamethasone at approximately 1 week intervals and will be determined at random by study staff.

The primary outcome for visits 2-3 will be to measure the effects of Ex-9 on fasting glucose-stimulated insulin secretion before and after experimentally induced insulin resistance. The primary experimental variable for analysis will be C-peptide during the clamp. Mean values will be compared between the period of glucose only stimulation and glucose with Ex-9. For each subject in the active treatment arm data will be analyzed using 2-way ANOVA for repeated measures using time (0-60 vs 60-120 min) and treatment (Dex vs no Dex) as the two factors. Based on the investigators' previous studies the investigators expect a significant time effect due to Ex-9. If there is an interaction with treatment the investigators would conclude that experimental insulin resistance influences the fasting GLP-1 effect. Data from control subjects will be analyzed identically; here the investigators expect no interaction, indicating that the fasting GLP-1 is a stable measure. In the investigators' previous study using Ex-9 during a glucose clamp, the average coefficient of variation in insulin concentrations at the conclusion of each step in the ramp was 30%. Using this estimate of between subject variation, detecting a 20% difference between subsequent steps in the GLP-1 ramp with a power of 80% and significance level of 0.05 will require 8 subjects.

AIM3: The purpose of Aim-3 of this study is to determine the role of basal GLP-1 action on fasting glucose regulation in lean, obese, pre-diabetic and type 2 diabetic (T2DM) subjects. Approximately 15-20 subjects will complete this cross sectional study of age-matched subjects across the spectrum of glucose tolerance will be used to test the hypothesis that fasting GLP-1 action increases as beta-cell function declines.

Enrolled participants for Aim-3 will be asked to complete two study visits including the consent visit and one infusion visit that will include a hyperglycemic clamp and an infusion of the antagonist Exendin (9-39). The infusion procedure will last approximately 2 hours.

The primary outcome measure for Aim-3 will be the fasting GLP-1 effect. This will be defined as the difference in steady state glucose-stimulated insulin secretion with and without Ex-9. The difference will be expressed as a percentage of glucose stimulated insulin secretion without Ex-9, and serve as the primary variable for comparison among the lean, obese and diabetic cohorts.

ELIGIBILITY:
Inclusion Criteria:

AIM2: SELECTION OF HEALTHY SUBJECTS

* Healthy adults age 20-45 years
* Body Mass Index (BMI) less than or equal to 35.0 kg/m2
* HbA1c less than or equal to 5.7% as measured at screening visit
* Ability to speak and understand English

AIM3: NON-DIABETIC SUBJECTS

* Adults age 18-65 years
* Body Mass Index (BMI) 25-40.0 kg/m2
* HbA1c less than or equal to 6.5% as measured at screening visit
* No Diabetes or use of diabetes medications such as insulin or metformin
* Ability to speak and understand English

AIM3: DIABETIC Type II SUBJECTS

* Adults age 18-65 years
* Body Mass Index (BMI) 25-40.0 kg/m2
* HbA1c less than or equal to 7.5% plus a diagnosis of Type II diabetes managed by either Metformin, Sulfonylurea, or diet and exercise
* Ability to speak and understand English

Exclusion Criteria:

AIM2:

* Uncontrolled high blood pressure
* Diabetes or use of diabetes medications such as insulin or metformin
* Evidence of active heart disease, unstable angina or heart failure
* Lung disease or COPD
* Malabsorptive GI disease, such as celiac disease, or gastric bypass
* Significant hepatic disease
* Kidney disease or renal insufficiency (eGFR < 60 mL/kg/min)
* Untreated anemia (hematocrit < 34%) as measured at screening visit
* Pregnant females
* Active substance abuse
* Chronic use of oral steroid medications such as prednisone and hydrocortisone
* Apparent sensitivity to any study peptides as determined by the skin test
* Diagnosis or h/o PTSD
* Active mental health disorders such as depression, or as a result of Traumatic Brain Injury (TBI)

AIM3: ALL SUBJECTS

* Uncontrolled high blood pressure
* Evidence of active heart disease, unstable angina or heart failure
* Lung disease or COPD
* Malabsorptive GI disease, such as celiac disease, or gastric bypass
* Significant hepatic disease
* Kidney disease or renal insufficiency (eGFR < 60 mL/kg/min)
* Untreated anemia (hematocrit < 34%) as measured at screening visit
* Pregnant females
* Active substance abuse
* Chronic use of oral steroid medications such as prednisone and hydrocortisone
* Apparent sensitivity to any study peptides as determined by the skin test
* Diagnosis or h/o PTSD
* Active mental health disorders such as depression, or as a result of Traumatic Brain Injury (TBI)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David D'Alessio, MD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Aim 3 not initiated, no participants enrolled in Aim 3 Arms/Groups
Period: Hyperglycemic Clamp + Exendin (9-39)
Arm/Group | Hyperglycemic Clamp + Exendin (9-39)
Started | 6
Completed | 6
Not Completed | 0
Period: With Dexamethasone
Arm/Group | Hyperglycemic Clamp + Exendin (9-39)
Started | 6
Completed | 5
Not Completed | 1
Not completed — No IV access | 1

BASELINE CHARACTERISTICS:
Groups:
- Hyperglycemic Clamp + Exendin (9-39): During the 2-hour procedure, a variable infusion of 20% dextrose and blood glucose will be clamped at basal + 3mM. Participants will receive an infusion of the GLP-1 receptor antagonist Exendin (9-39) between the 60-120 minute time-points of the clamp. The amount of Ex-9 infused will be 750 pmol/kg/min for 60 minutes.
  Exendin (9-39): Upon establishing a hyperglycemic clamp (target blood glucose at basal +3 mM) Exendin (9-39) will be infused.
  Hyperglycemic Clamp: A variable infusion of 20% dextrose will begin to clamp the blood glucose at basal +3 mM.
  Each subject then received dexamethasone 4 mg daily for 7 days and returned for an identical experiment with a hyperglycemic clamp and exendin-(9-39).
Arm/Group | Hyperglycemic Clamp + Exendin (9-39)
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: AIM2: C-peptide Levels.
Description: Primary variable for analysis will be C-peptide during the clamp. Mean values will be compared between the control and dexamethasone studies for C-peptide levels during the hyperglycemia plus exendin-(9-39) period of the clamps. For each subject the mean C-peptide during the 60-90 minute period of the initial study (with no dexamethasone) will be compared to the 60-120 period with dexamethasone.
Time Frame: Minute infusion periods (0-60 vs 60-120) baseline and treatment (Dex vs no Dex)
Population: Data not collected for one subject
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Hyperglycemic Clamp + Exendin (9-39)
Number analyzed (Participants) | 5
ng/ml
  Control + exendin-(9-39) | 10,335 (1984)
  Dexamethasone + exendin-(9-39) | 9042 (1255)

2. Primary Outcome: AIM3: To Determine the Fasting GLP-1 Effect.
Description: The fasting GLP-1 effect will be defined as the difference in steady state glucose stimulated insulin secretion with and without Ex-9.
Time Frame: Minute infusion periods (0-60 vs 60-120)
Population: Data not collected
Arm/Group | Hyperglycemic Clamp + Exendin (9-39)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 weeks
Groups:
- Hyperglycemic Clamp + Exendin (9-39) With Dexamethasone; Hyperglycemic Clamp + Exendin (9-39) Without Dexamethasone: During the 2-hour procedure, a variable infusion of 20% dextrose and blood glucose will be clamped at basal + 3mM. Participants will receive an infusion of the GLP-1 receptor antagonist Exendin (9-39) between the 60-120 minute time-points of the clamp. The amount of Ex-9 infused will be 750 pmol/kg/min for 60 minutes.
  Exendin (9-39): Upon establishing a hyperglycemic clamp (target blood glucose at basal +3 mM) Exendin (9-39) will be infused.
  Hyperglycemic Clamp: A variable infusion of 20% dextrose will begin to clamp the blood glucose at basal +3 mM.
  Each subject then received dexamethasone 4 mg daily for 7 days and returned for an identical experiment with a hyperglycemic clamp and exendin-(9-39).
  The study protocol and exposures were identical for each subject on the 1 (six subjects) or 2 (five subjects) days they were studied, and differed only by preceding dexamethasone treatment (5 subjects). Other Adverse Events are reported above separately for the experiments with and without dexamethasone.
Arm/Group | Hyperglycemic Clamp + Exendin (9-39) With Dexamethasone | Hyperglycemic Clamp + Exendin (9-39) Without Dexamethasone
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/6 | 5/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hyperglycemic Clamp + Exendin (9-39) With Dexamethasone (N=6) | Hyperglycemic Clamp + Exendin (9-39) Without Dexamethasone (N=6)
Bruising at IV site (General disorders) | 3 (3) | 0 (0)
Transient Nausea (General disorders) | 1 (1) | 1 (1)
Dizziness (General disorders) | 0 (0) | 2 (2)
Blood glucose levels between 70 and 80 mg/dl that were asymptomatic (General disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Difficulty recruiting healthy veterans who were established at the Durham VA for this study. Healthy subjects were not frequently enrolled with VA healthcare and veterans enrolled with the VA did not often meet the inclusion/exclusion criteria.

Enrollment was also limited by the COVID-19 pandemic.

Due to the small sample with collected data statistical analysis was not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-18): https://cdn.clinicaltrials.gov/large-docs/07/NCT02844907/Prot_SAP_000.pdf